CLINICAL TRIAL: NCT03220971
Title: Theranostic Translation Applications Against Viral, Metabolic Liver Diseases and Hepatic Oncogenesis: Lipoprotein and Apolipoproteins at a Crossroad
Brief Title: Lipoprotein and Apolipoproteins With Metabolic Liver Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chun-Hsiang Wang (Other)
Responsible Party: Sponsor-Investigator, Chun-Hsiang Wang, Tainan Municipal Hospital, Tainan Municipal Hospital
Organization: Tainan Municipal Hospital (Other)
Other Study IDs: 1060603
Record Dates: First submitted 2017-07-03; First posted 2017-07-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Disorders of Lipoprotein Metabolism and Other Lipidaemias
Keywords: Lipoprotein and Apolipoproteins metabolism
MeSH Terms: interventions — Lipoproteins; Apolipoproteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biochemical blood: GOT, GPT, HDL, LDL, TG, insulin, AC sugar
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- proposed cross-section study: 1. 100 subjects with NAFLD/NASH and negative anti-HCV Ab
  2. 50 subjects with HCC and negative anti-HCV Ab
  3. 50 subjects with HCC and positive for genotype-1 HCV
  4. 50 controls with all negative for NAFLD/NASH but positive for genotype-1 HCV
  5. 50 controls with all negative for NAFL, NASH and HCV
  Interventions: Other: lipoprotein and apolipoproteins
- proposed longitudinal study: 1. 50 NAFLD/NASH patients and positive for genotype-1 HCV with SVR
  2. 10 NAFLD/NASH patients and positive for genotype-1 HCV without SVR
  3. 10 HCC patients and positive for genotype-1 HCV with SVR
  4. 10 HCC patients and positive for genotype-1 HCV without SVR
  5. 50 chronic hepatitis C but not NAFLD patients with SVR
  6. 10 chronic hepatitis C but not NAFLD patients without SVR
  Interventions: Other: lipoprotein and apolipoproteins

INTERVENTIONS:
Other: lipoprotein and apolipoproteins — To find out the role of lipoprotein and apolipoproteins (apos) in pathogenic hepatic diseases

SUMMARY:
Theranostic translation applications against viral, metabolic liver diseases and hepatic oncogenesis: lipoprotein and apolipoproteins at a crossroad

DETAILED DESCRIPTION:
An intimate link between microbial infections, metabolic changes and oncogenesis has been drawn attentions increasingly, indicating a crossroad leading to pathogenesis and disease progression. Globally the burden of hepatitis B and C virus infections is 450 and 185 millions, respectively and chronic hepatitis disease causes a high risk of liver cirrhosis, hepatocellular carcinoma and metabolic disorders

ELIGIBILITY:
Inclusion Criteria:

1. above 20 years
2. nonalcoholic fatty liver disease
3. Non-Alcoholic Steatohepatitis

Exclusion Criteria:

1. alcohonic hepatitis 2. Autoimmune liver disease 3. HIV postive

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An intimate link between microbial infections, metabolic changes and oncogenesis has been drawn attentions increasingly, indicating a crossroad leading to pathogenesis and disease progression. Globally the burden of hepatitis B and C virus infections is 450 and 185 millions, respectively and chronic hepatitis disease causes a high risk of liver cirrhosis, hepatocellular carcinoma and metabolic disorders
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Theranostic Translation Applications Against Viral, Metabolic Liver Diseases and Hepatic Oncogenesis: Lipoprotein and Apolipoproteins at a Crossroad | 2years
  Study the interplay between hepatitis C virus (HCV) and lipid metabolism(the HCV infection affects host lipid homeostasis, regarding transportation, synthesis, and catabolism.)

CONTACTS AND LOCATIONS:
Locations (1):
- Chun-Hsiang Wang, Tainan, Taiwan